CLINICAL TRIAL: NCT06486649
Title: Application of a Multimodal Large Language Model to Assist Diagnosis for Heart Failure With Preserved Ejection Fraction
Brief Title: Application of Multimodal Large Language Model in HFpEF
Acronym: MeG-HFpEF
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); The First Hospital of Hebei Medical University (Other); Qianfoshan Hospital (Other); Qingdao Municipal Hospital (Other)
Responsible Party: Principal Investigator, Tang Yida, Professor, Peking University Third Hospital
Other Study IDs: M2023830
Record Dates: First submitted 2023-12-22; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: Heart failure with preserved ejection fraction; large language model; diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single group: The routine consultation process was performed first: according to the process recommended by the 2023 edition of the Chinese Expert Consensus on the Diagnosis and Treatment of Heart Failure with Preserved Ejection Fraction, the attending cardiologist completed the subject's clinical criteria assessment and performed the HFpEF diagnosis (yes/no).
  During the attending physician's checkup visit, the multimodal large language model screening system (MedGuide-72B) collected routine visit data, recorded relevant data and indicators during the patient's communication with MedGuide-72B and made the diagnosis.
  Interventions: Diagnostic Test: Multimodal Large Language Model Diagnosis; Diagnostic Test: Routine diagnostic and therapeutic procedure

INTERVENTIONS:
Diagnostic Test: Multimodal Large Language Model Diagnosis — Diagnosis for heart failure with preserved ejection fraction (HFpEF) using the multimodal large language model MedGuide-72B.
Diagnostic Test: Routine diagnostic and therapeutic procedure — Routine diagnostic and therapeutic procedure

SUMMARY:
This study will validate the effectiveness of a multimodal large language model to screen for heart failure with preserved ejection fraction (HFpEF), comparing it with the traditional clinical standardized assessment process.

DETAILED DESCRIPTION:
Heart failure is a major complication of various heart diseases and is the leading lethal cause of cardiovascular death worldwide. Based on the left ventricular ejection fraction (LVEF), heart failure can be divided into heart failure with reduced ejection fraction (HFrEF), heart failure with preserved ejection fraction (HFpEF) and heart failure with mildly reduced ejection fraction (HFmrEF). Heart failure rehospitalization rates and in-hospital complications did not differ between HFrEF and HFpEF. However, over the past two decades, the survival rate of HFrEF has improved significantly, whereas HFpEF has remained stagnant. One of the major reasons for this is that the diagnostic process of HFpEF is complicated, and it is easy to cause missed diagnosis in the clinic, resulting in delayed treatment.

Multimodal large language models are capable of integrating and analyzing medical data from different sources, including textual data (e.g., medical records, medical literature), image data (e.g., electrocardiograms, CT scan images), and audio data (e.g., symptoms narrated by patients). This multimodal data integration capability is crucial for understanding complex medical scenarios, as it provides a more comprehensive view of the condition than a single data source.

The diagnosis of HFpEF faces many challenges and requires clinicians to make judgments on multi-dimensional data, which can easily lead to the underdiagnosis and misdiagnosis of the disease. As a generative artificial intelligence tool, a large language model is able to integrate and analyze data from different sources and has the ability to learn and evolve from existing clinical evidence. Based on this, this study intends to evaluate the effectiveness of multimodal large language model for screening for heart failure with preserved ejection fraction (HFpEF), comparing it with the traditional clinical standard assessment process.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or female;
2. Cardiology inpatients with suspected heart failure with preserved ejection fraction (cardiac ultrasound suggestive of LVEF ≥50% with at least 1 of the following: 1, left ventricular hypertrophy and/or left atrial enlargement; and 2, abnormal diastolic cardiac function);
3. Current or previous at least one symptom of heart failure, including dyspnea (including exertional dyspnea, nocturnal paroxysmal dyspnea, and telangiectasia), malaise, nausea, and bilateral lower extremity edema;
4. Voluntary participation and signed informed consent.

Exclusion Criteria:

1. Acute heart failure or acute worsening of chronic heart failure;
2. Severe coronary stenosis (≥75% stenosis) without revascularization;
3. Patients who are unable to perform exercise stress echocardiography or have contraindications to the test;
4. are participating in other clinical trials;
5. Those with severe organic pathologies of the liver, kidney, or hematologic system or those with chronic diseases;
6. Those who are unable to follow the trial procedures;
7. Those who refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients routinely hospitalized in the cardiology department who also met the needs of this trial and are not recruited separately.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
dignostic specificity | through study completion, an average of 8 months
  dianostic specificity comparison between routine diagnosis and therapy and large language model diagnosis
dignostic sensitivity | through study completion, an average of 8 months
  dianostic sensitivity comparison between routine diagnosis and therapy and large language model diagnosis

SECONDARY OUTCOMES:
consistency rate | through study completion, an average of 8 months
  consistency rate between routine diagnosis and therapy and large language model diagnosis
time spent on diagnosis | through study completion, an average of 8 months
  comparison of time spent on diagnosis between routine diagnosis and therapy and large language model diagnosis
patient satisfaction | through study completion, an average of 8 months
  comparison of patient satisfaction between routine diagnosis and therapy and large language model diagnosis by questionnaire
economic cost analysis | through study completion, an average of 8 months
  comparison of economic cost between routine diagnosis and therapy and large language model diagnosis by the total cost of treatment
false discovery rate | through study completion, an average of 8 months
  comparison of false discovery rate between routine diagnosis and therapy and large language model diagnosis
physician workload assessment | through study completion, an average of 8 months
  comparison of physician workload between routine diagnosis and therapy and large language model diagnosis according to counting the number of participants with treatment-related
diagnosis efficiency | through study completion, an average of 8 months
  The probability of accuracy compared to the final diagnosis of the patient's visit

CONTACTS AND LOCATIONS:
Locations (1):
- Peking UniversityThird Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kittleson MM, Panjrath GS, Amancherla K, Davis LL, Deswal A, Dixon DL, Januzzi JL Jr, Yancy CW. 2023 ACC Expert Consensus Decision Pathway on Management of Heart Failure With Preserved Ejection Fraction: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2023 May 9;81(18):1835-1878. doi: 10.1016/j.jacc.2023.03.393. Epub 2023 Apr 19. No abstract available. PMID 37137593
- [Background] Wang X, Cunningham JW. Restoring balance in heart failure with preserved ejection fraction. Eur J Heart Fail. 2022 Aug;24(8):1415-1417. doi: 10.1002/ejhf.2599. Epub 2022 Jul 18. No abstract available. PMID 35789069
- [Background] Sicari R. Phenotyping heart failure with preserved ejection fraction with exercise stress echocardiography. Eur Heart J Cardiovasc Imaging. 2022 Jul 21;23(8):1053-1054. doi: 10.1093/ehjci/jeac053. No abstract available. PMID 35262693
- [Background] Omote K, Verbrugge FH, Borlaug BA. Heart Failure with Preserved Ejection Fraction: Mechanisms and Treatment Strategies. Annu Rev Med. 2022 Jan 27;73:321-337. doi: 10.1146/annurev-med-042220-022745. Epub 2021 Aug 11. PMID 34379445
- [Background] Margulies KB. DELIVERing Progress in Heart Failure with Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1138-1140. doi: 10.1056/NEJMe2210177. Epub 2022 Aug 27. No abstract available. PMID 36027566
- [Background] Ventura HO, Lavie CJ, Mehra MR. Heart Failure With Preserved Ejection Fraction: Separating the Wheat From the Chaff. J Am Coll Cardiol. 2020 Jan 28;75(3):255-257. doi: 10.1016/j.jacc.2019.11.027. No abstract available. PMID 31976862
- [Background] Reddy YNV, Borlaug BA. Heart Failure With Preserved Ejection Fraction: Where Do We Stand? Mayo Clin Proc. 2020 Apr;95(4):629-631. doi: 10.1016/j.mayocp.2020.02.015. No abstract available. PMID 32247333
- [Background] Donal E, L'official G, Kosmala W. Heart Failure With Preserved Ejection Fraction: Defining Phenotypes. J Card Fail. 2020 Nov;26(11):929-931. doi: 10.1016/j.cardfail.2020.09.013. Epub 2020 Sep 19. No abstract available. PMID 32956811
- [Background] Ahmad T, Desai NR, Januzzi JL. Heart Failure With Preserved Ejection Fraction: Many Emperors With Many Clothes. JACC Heart Fail. 2020 Mar;8(3):185-187. doi: 10.1016/j.jchf.2019.11.004. Epub 2020 Jan 8. No abstract available. PMID 31926855